CLINICAL TRIAL: NCT04774289
Title: Incidence of Malignant Peripheral Nerve Sheath Tumors Development in Patients With Neurofibromatosis Type 1 Receiving and Not Receiving Medical Therapies Directed at Plexiform Neurofibromas
Brief Title: Incidence of Malignant Peripheral Nerve Sheath Tumor (MPNST) Development in Participants With Neurofibromatosis Type 1 (NF1) Receiving and Not Receiving Medical Therapies Directed at Plexiform Neurofibromas (PN)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000271; 000271-C
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06-24

CONDITIONS: Neurofibromatosis 1; Peripheral Nerve Neoplasms, Malignant
Keywords: Retrospective Review; Natural History; genetic tumor predisposition syndrome
MeSH Terms: conditions — Neurofibromatosis 1; Peripheral Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants with NF1 seen at the NIH from 1/1/1998 to 1/1/2020

SUMMARY:
Background:

NF1 is a genetic syndrome. Tumors appear early in life. Many people with NF1 develop PN. These tumors can become an aggressive cancer called MPNST. People with MPNST may benefit from treatment with a MEK inhibitor (MEKi). Researchers want to learn if there is an increased risk of MPNST formation from MEKi treatment in people with NF1. To do this, they will review data that has been collected in NIH NF1 studies.

Objective:

To describe the characteristics of people who have taken part in NF1 studies at NIH and to compare the risk of MPNST formation in those treated with MEKi or other PN-directed treatment.

Eligibility:

People with NF1 who were seen at NIH from Jan. 1, 1998, to Jan. 1, 2020.

Design:

Participants medical records will be reviewed. Participants who opted out of future use of their data will not be included.

Demographic data, like sex, race, and date of birth, will be collected.

Data about MEKi and non-MEKi treatments will be collected.

Clinical data, such as surgery and treatment details, will be collected.

The differences between all participants who were seen at NIH for any NF1 related study will be compared. Participants will be put into 4 groups:

History of MEKi therapy

Treatment with tumor directed therapy other than MEKi

Treatment with both MEKi and non-MEKi tumor directed therapies

No tumor directed medical therapy

Participants with NF1 who were treated for PN with either a MEKi treatment or a non-MEKi treatment will also be compared.

The study will last for 3 to 6 months.

DETAILED DESCRIPTION:
Study Description: This is a retrospective review that includes all patients with NF1 enrolled on natural history and treatment trials at the National Cancer Institute (NCI) from 1/1/1998 to 1/1/2020, excluding patients referred for treatment of MPNST.

Objective: To describe the clinical and demographic characteristics of NF1 study participants who come for evaluation at the NCI and to compare the risk of MPNST formation in patients treated with MEK 1/2 inhibitor (MEKi) or other PN-directed treatment.

Study Population: All participants with NF1 seen at the NIH from 1/1/1998 to 1/1/2020

Description of Sites/Facilities conducting research: This is a single site study initiated by the Pediatric Oncology Branch at the National Cancer Institute

Study Duration: Data abstraction to completion of data analyses will take 3-6 months.

ELIGIBILITY:
* Inclusion Criteria:
* All participants seen at the NIH from 1/1/1998 to 1/1/2020 with a clinical or laboratory diagnosis of NF1
* Participants beyond the neonatal period (4 weeks).

Exclusion Criteria:

-All participants seen at the NIH from 1/1/1998 to 1/1/2020 with a clinical or laboratory diagnosis of NF1 who opted out of future use.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
risk of MPNST formation | ongoing
  descriptive statistics and frequency distribution of selected variables

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States